CLINICAL TRIAL: NCT05993143
Title: A Multicentre, Phase III, Double-blind, Randomised, Parallel, Placebo-controlled Trial to Assess Efficacy and Safety of Early Administration of Ivermectin During 3 Consecutive Days to Prevent SARS CoV-2 (COVID-19) Hospitalisation in Adults Older Than 50 Years of Age
Brief Title: Ivermectin to Prevent SARS-CoV-2 (COVID-19) Hospitalisation in Subjects Over 50
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped because no statistically significant difference was observed in the interim analysis. With high vaccine rates in those over 50 and an expected low incidence, it would not be feasible to complete recruitment within a short period.
Sponsor: Insud Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVER-303
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: ivermectin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Test (Ivermectin) and reference (placebo) tablets will be identical in size, colour, taste and appearance. The packaging and labelling will not allow for any distinction between the test and reference drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (test product) (Experimental): Ivermectin 9 mg and 18 mg immediate-released tablets to be taken orally once daily during 3 days at 600 µg/kg/day ± 120 µg/kg/day depending on their body weight.
  Interventions: Drug: Ivermectin
- Placebo (reference product) (Placebo Comparator): Placebo tablets to be taken orally once daily during 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — Round and white tablets
  Other Names: Ivermectin 9 mg and 18 mg
  Arms: Ivermectin (test product)
Drug: Placebo — Round and white tablets
  Arms: Placebo (reference product)

SUMMARY:
The primary objective of this study is to assess the efficacy of early administration of ivermectin for three consecutive days to prevent SARS-CoV-2 hospitalisation in adults older than 50 years of age. Secondary objectives include assessing the efficacy of an early administration of ivermectin for three consecutive days to prevent SARS-CoV-2 disease progression in adults older than 50 years of age and evaluating the safety and tolerability of ivermectin in SARS-CoV-2 infected adults older than 50 years of age.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, multicentre trial in parallel groups. During the screening/enrollment phase (Visit 1.1 to Visit 1.3) informed consent will be obtained and the screening procedures will be performed. A rapid antigen-based test will be offered to all patients who do not have a polymerase chain reaction (PCR) or a rapid antigen-based test result at screening (each of these tests may be considered a part of the standard procedure of the site). Eligible subjects will be randomised 1:1 to receive ivermectin or placebo. The subjects will be dispensed investigational product (IP), based on their body weight, and will take the first dose of IP at site. The subjects will receive portable pulse oximeters for peripheral capillary oxygen saturation (SpO2) monitoring at home. The treatment phase will last 3 days and include an on-site Visit 1.3 and phone call Visits 2 and 3 which will be performed on the following 2 days. PCR test or rapid antigen test results will be communicated to subjects as soon as available. Subjects with negative COVID-19 PCR test or rapid antigen test results will be withdrawn from the trial unless they have a positive rapid antigen test or COVID-19 PCR test result a few days later. The subjects will be followed up until Day 28.

During the follow-up, the subjects will have phone call Visits 4 to 9 every other day, followed by Visit 10 after one week (Day 21). The subjects will be asked to measure oxygen saturation as well as body temperature during all phone call visits and report the respective results to the investigator. The on-site Visit 11 is the last visit (Day 28). The subjects will return IPs (including empty and partially empty containers) and pulse oximeters.

In addition, the subjects will be provided with a contact number available 24/7 to contact the investigator if their condition worsens. In case of health condition worsening (dyspnoea, fever [body temperature ≥ 37.8°C] lasting for more than 6 days, SpO2 ≤ 95% or any other worsening criteria based on the investigator's judgement) confirmed during the phone call visit, the subjects will have an unscheduled visit at the site.

The subjects will be hospitalised if they fulfill any of the following criteria: pneumonia confirmed by chest X-ray; SpO2 ≤ 94% or partial pressure of oxygen in blood (PO2) < 80 mmHg in gasometry; respiratory frequency > 20 rpm; fever (body temperature ≥ 37.8°C) for more than 6 days plus one of the following analytic parameters: C-reactive protein (CRP) > 5 mg/dL, ferritin > 500 ng/mL or D dimer > 700 ng/mL. If there is any other condition that requires hospitalisation as per investigator judgement, the condition has to be documented in detail in the subject's file including a description whether the hospitalisation was performed due to SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult > 50 years of age
2. SARS-CoV-2 infection diagnosed either through a rapid antigen-based test or an RNA based reverse-transcription polymerase chain reaction (RT-PCR) diagnostic test performed in nasopharyngeal sample
3. Onset of COVID-19 symptoms < 120 hours (5 days) prior to screening
4. Written informed consent
5. For females of childbearing potential only: They must declare that they did not intend to become pregnant in the last month prior to screening and they do not intend to become pregnant for one month following the last IP administration. For males who have partners of childbearing potential: Willing to use condoms until 3 months after last IP intake.
6. Negative result for urine pregnancy test (women of childbearing potential only)

Exclusion Criteria:

1. Intake of Ivermectin within 30 days before screening
2. Routine intake of antivirals, including antiretroviral treatment
3. Allergy, hypersensitivity or contraindication to Ivermectin, metabolites or excipients
4. Subjects with symptoms of disease severity (dyspnoea, SpO2 ≤ 94%)
5. Subjects requiring hospitalisation for any reason.
6. Epidemiological risk or suspicion of being infected by Loa loa or other filariases
7. Previous enrolment in this trial or participation in any other drug investigational trial within the past 30 days (or five half-lives of IP whichever is longer) prior to screening
8. Weight < 50 kg
9. Pregnancy or lactation
10. Inability to take oral medications
11. At least one of the following acute/chronic disease or deficiency:

    1. History of bone marrow transplant or haematopoietic systems diseases
    2. Moderate or severe liver disease (Child Pugh score ≥ B or ALT [alanine transaminase] or AST [aspartate transaminase] > 3 times upper limit as determined at screening visit), severe cholestasis, cirrhosis or severe hepatic failure
    3. Transplanted patient under immunosuppressive treatment, disease that may need immunosuppressive treatments or other medical conditions that under the judgement of investigator would not benefit the patient to be included (including but not limited to psoriasis, G6PD (glucose-6-phosphate dehydrogenase) deficiency, porphyria, history of diverticulosis, seizure disorder, concurrent malignancy requiring chemotherapy, ongoing skin infection (e.g. pyodermitis) or evidence of current tuberculosis including latent untreated tuberculosis)
    4. Ophthalmological or recent/ongoing neurological diseases
12. Active cardiac disease or a history of cardiac dysfunction including any of the following:

    1. History of angina pectoris, symptomatic pericarditis, or myocardial infarction within 12 months prior to screening
    2. History of congestive heart failure (New York Heart Association functional classification III-IV)
13. Concomitant use of barbiturates, sodium oxybate, valproic acid or warfarin
14. Laboratory abnormalities relevant for the trial, including but not limited to: neutropenia < 500/mm3, thrombocytopenia < 100,000/mm3
15. Any other significant disease, disorder or finding which, in the opinion of the investigator, may significantly increase the risk to the subject because of participation in the study, affect the ability of the subject to participate in the study or impair interpretation of the study data
16. Employees of the investigator or clinical trial site, with direct involvement in the proposed trial or other studies under the direction of that investigator or clinical trial site, as well as family members of the employees or the principal investigator
17. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Hospitalisation due to SARS-CoV-2 | day 1 to day 28
  Percentage of subjects requiring SARS-CoV-2 hospitalisation during 28 days after first IP administration.

SECONDARY OUTCOMES:
Change in subjects' clinical status | day 1, 2, 3, 4, 6, 8, 10, 12, 14, 21 and 28
  Efficacy of an early administration of Ivermectin for three consecutive days to prevent SARS-CoV-2 disease progression in adults older than 50 years of age.
Occurrence of any adverse event related to Ivermectin treatment | day 1, 2, 3, 4, 6, 8, 10, 12, 14, 21 and 28
  Evaluation of safety and tolerability of Ivermectin in SARS CoV 2 infected adults older than 50 years of age

CONTACTS AND LOCATIONS:
Locations (20):
- Spain (20):
  - Hospital de Poniente, El Ejido, Almeria
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital San Pedro, Logroño, La Rioja
  - HM Montepríncipe, Boadilla del Monte, Madrid
  - HM Puerta del Sur, Móstoles, Madrid
  - HM Torrelodones, Torrelodones, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario A Coruña-CHUAC, A Coruña
  - Centro de Atención Primaria Les Corts, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid
  - HM Sanchinarro, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No